CLINICAL TRIAL: NCT00637845
Title: A Multi-centred, Phase IV, Post-Marketing, Prospective, Randomized, Double-Blind Study Comparing Esomeprazole Magnesium 40mg Once Daily Versus Lansoprazole 30 mg Twice Daily in Symptom Control of Subjects With Persistent Gastrooesophageal Reflux Disease While on 30mg Once Daily Lansoprazole Therapy
Brief Title: Study Comparing Esomeprazole Magnesium 40mg Once Daily Versus Lansoprazole 30 mg Twice Daily in Symptom Control of Subjects With Persistent Gastrooesophageal Reflux Disease (GERD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Tore Lind, MD - Nexium Medical Science Director, Astra Zeneca
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 311; D9612L00055 (Other: AZ)
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Heartburn; Gastroesophageal Reflux Disease
Keywords: Nexium; Esomeprazole Magnesium; Gastroesophageal Reflux Disease; Heartburn
MeSH Terms: conditions — Heartburn; Gastroesophageal Reflux | interventions — Esomeprazole; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): 40mg once daily
  Interventions: Drug: Esomeprazole Magnesium
- 2 (Active Comparator): 30mg twice daily
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Esomeprazole Magnesium — 40mg once daily
  Other Names: Nexium
  Arms: 1
Drug: Lansoprazole — 30mg twice daily
  Other Names: Prevacid
  Arms: 2

SUMMARY:
A double-blind study comparing Esomeprazole Magnesium 40 mg once daily and Lansoprazole 30 mg twice daily to control the symptoms in patients with gastroesophageal reflux disease (GERD) with continued heartburn symptoms with a course of therapy of 30 mg twice daily Lansoprazole.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have reported history of heartburn symptoms whilst on lansoprazole 30 mg twice daily during the 30 days prior to screening.
* Subjects must have a minimal cumulative heartburn score of at least 4 for a minimum of 14 days, where zero = none, one = mild, two = moderate, three = severe.

Exclusion Criteria:

* subjects history of esophageal ulcers, esophageal strictures, esophageal neoplasms, gastric or duodenal ulcers, or any other significant gastric or esophageal pathology judged to be clinically significant by the investigator.
* Subjects with persistent heartburn symptoms while on lansoprazole 30 mg twice daily for a period of > 6 months
* Subjects with a history of severe hepatic insufficiency (specifically, Childs-Pugh Class C liver disease) that may adversely affect the metabolism abd pharmacokinetics of esomeprazole and/or lansoprazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2002-06; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
To compare the clinical efficacy of esomeprazole magnesium 40mg once daily versus lansoprazole 30 mg twice daily in symptom control of heartburn in subjects with heartburn symptoms resistant to 30 mg once daily therapy of lansoprazole. | Heartburn symptoms collected on diary card daily

SECONDARY OUTCOMES:
To compare efficacy of esomeprazole magnesium 40mg daily vs lansoprazole 30 mg twice daily in symptom control of acid regurgitation, epigastric pain, and night-time heartburn in subjects with GERD symptoms resistant to 30 mg daily therapy of lansoprazole | Heartburn symptoms collected on diary card daily
To evaluate the use of supplementary antacids (as heartburn rescue therapy) in subjects treated with esomeprazole magnesium 40 mg once daily versus lansoprazole 30 mg twice daily | Heartburn symptoms collected on diary card daily
To assess tolerability of esomeprazole magnesium 40 mg twice daily versus lansoprazole 30 mg twice daily. | Ongoing Adverse event collection

CONTACTS AND LOCATIONS:
Overall Officials: Paula Fernstrom, Study Director — Nexium Global Product Director, AstraZeneca